CLINICAL TRIAL: NCT03827603
Title: Ibrutinib in Steroid Refractory Autoimmune Hemolytic Anemia: ELaboration of Treatment Approach
Brief Title: Ibrutinib in Steroid Refractory Autoimmune Hemolytic Anemia
Acronym: ISRAEL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eugene Nikitin (Other)
Responsible Party: Sponsor-Investigator, Eugene Nikitin, Professor, Association of Oncological Hematologists
Organization: Association of Oncological Hematologists (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54179060CLL2013
Record Dates: First submitted 2019-01-24; First posted 2019-02-01 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: AIHA - Warm Autoimmune Hemolytic Anemia
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with AIHA and CLL (Experimental): patients with CLL and in Steroid Refractory AIHA receive ibrutinib 420 mg per day till progression or intolerance
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib and rituximab combination for the treatment of steroid refractory AIC (warm type AIHA and PRCA) with underlying CLL.
  Other Names: Imbruvica

SUMMARY:
This is an open-labeled, single arm, Phase II, two staged study of combination of ibrutinib and rituximab in patients with autoimmune cytopenia and underlying CLL. In stage I (remission induction) patients will receive ibrutinib and rituximab for 6 months; in stage II (maintenance) - only ibrutinib until relapse, progression or unacceptable toxicity. A total of 50 patients will be enrolled into the trial. The results will be compared to historical control, efficacy of rituximab as monotherapy or in combination with chemotherapy in patients with AIC and underlying CLL.

DETAILED DESCRIPTION:
Subjects will give informed consent before any protocol specific assessments. Blood samples, physical examination, CT scan and bone marrow examination will be performed to determine baseline disease status and study eligibility. All examinations must be performed ≤ 14 days prior to first infusion, with the exception of the CT scan and bone marrow examination. The CT scan and the bone marrow examination will be performed within 6 weeks of first infusion.

treatment regimen: Rituximab 375 mg/m2 8 weekly infusions (days 1, 8, 15, 22, 29, 36, 43, 50, 57), then 3 infusion every 28 days (days 85, 113, 141) Ibrutinib 420 mg (3 tablets) daily, constantly for 6 months

Disease status assessments to determine subject response or progression will be performed monthly according to NCI Criteria and will include:

* Physical examination including lymph node examination, spleen and liver measurement, and detection of constitutional symptoms
* Peripheral blood sample evaluation of complete blood count (CBC) and differential (expressed in % and absolutes)
* Direct antiglobulin test
* In addition, subjects will be monitored for safety, efficacy.

After completion of the induction phase, subjects achieving CR or PR (for AIC and CLL) will continue maintenance phase. During maintenance phase patients will receive:

ibrutinib 420 mg (3 tablets) daily, constantly until progression or unacceptable toxicity Survival and disease status assessments will be performed 1 month post treatment and every 2 months until total observation time.

In addition, subjects will be monitored for safety and efficacy.

* Bone marrow examination is required for confirmation of CR 1 months post final rituximab infusion. Minimal Residual Disease (MRD) assessment of the bone marrow aspirate will also be performed for subjects demonstrating a CR.
* In PRCA patients with clinical evidence of response for anemia the bone marrow examination is required independently of CLL status at 1 month post last rituximab infusion.
* All subjects with clinical CR will receive MRD assessment of the peripheral blood during maintenance phase. In subjects achieved MRD-negative result in blood in two consecutive measurements bone marrow examination is required for confirmation of CR.
* CT-Scans will be performed for patients achieving a CR, PR or SD at 1 month post last rituximab infusion. CT-Scans must be repeated every 12 months beginning since final assessment of response after induction phase.

Follow-up assessment for subjects experiencing CLL progression or relapse of AIC during the maintenance phase requires a 1 month post-treatment safety assessment. Subsequent follow up visits include assessment of survival status, date of next CLL therapy, type of therapy and response to therapy.

ELIGIBILITY:
Inclusion Criteria

1. Flow cytometry confirmation of immunophenotype with CD5, CD19, CD20, CD23, CD79b, and surface Ig prior to Visit 2
2. Proven diagnosis autoimmune hemolytic anemia or pure red cell aplasia
3. Relapse of AIHA/PRCA after steroids, splenectomy or rituximab or refractoriness to glucocorticosteroid hormones
4. No more than 2 lines of antileukemia treatment
5. Hematology values must be within the following limits:

   1. Absolute neutrophil count 1000/mm3 independent of growth factor support
   2. Platelets 100.000/mm3 or 50.000/mm3 if bone marrow involvement independent of transfusion support in either situation
6. Biochemical values within the following limits:

   1. Alanine aminotransferase and aspartate aminotransferase less 3 upper limit of normal (ULN)
   2. Total bilirubin less 1.5x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
   3. Serum creatinine less 2 x ULN or estimated Glomerular Filtration Rate more 40 mL/min/1.73 m2
7. Age ≥ 18 years
8. ECOG Performance Status of 0-2
9. Life expectancy of at least 6 months
10. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
11. Women who are pregnant or breastfeeding are ineligible for this study.
12. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 month after treatment
  Response rate defined by transfusion independence, hemoglobin level, DAT and duration of response of autoimmunity (DR-AI), defined as the interval between time point of best response and relapse of AIC. Relapses of CLL will be censored.

CONTACTS AND LOCATIONS:
Locations (1):
- Eugene Nikitin, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No